CLINICAL TRIAL: NCT00121524
Title: Effects of Epinephrine and I.V. Needle on CPR Outcome
Brief Title: Effects of Epinephrine and Intravenous (I.V.) Needle on Cardiopulmonary Resuscitation (CPR) Outcome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Petter Andreas Steen (Other)
Collaborators: Laerdal Medical (Industry); Ullevaal University Hospital (Other); Health Region East, Norway (Other); Norwegian Air Ambulance Foundation (Other); University of Oslo (Other)
Responsible Party: Sponsor-Investigator, Petter Andreas Steen, Professor Acute Medicine, University of Oslo
Organization: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 525-02201
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; resuscitation; epinephrine; intravenous; survival
MeSH Terms: conditions — Heart Arrest | interventions — Epinephrine; Atropine; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV yes (Experimental): Intravenous needle Epinephrine q 3 min during CPR Atropine 3 mg in initial asystole Amiodarone 300 mg iv after repeated failed defibrillation attempts
  Interventions: Drug: Epinephrine; Device: Intravenous needle; Drug: Atropine; Drug: Amiodarone
- IV no (No Intervention): The patient will not have an intravenous needle placed or given any drugs during CPR. If patient obtains spontaneous circulation, an intravenous needle is placed and patient can receive any drugs that are appropriate during the following treatment.

INTERVENTIONS:
Drug: Epinephrine — Epinephrine 1 mg is given iv. every 3 min during CPR
  Other Names: Adrenaline
  Arms: IV yes
Device: Intravenous needle — An intravenous needle in placed as soon as possible during CPR
  Arms: IV yes
Drug: Atropine — Atropine 3 mg iv in initial systole
  Other Names: Atropine sulfate
  Arms: IV yes
Drug: Amiodarone — amiodarone 300 mg iv after repeated failed defibrillation attempts
  Other Names: Amiodaron
  Arms: IV yes

SUMMARY:
Intravenous epinephrine has been part of the guidelines for cardiopulmonary resuscitation since the start. It improves outcome in animal studies, but has never been investigated in a controlled study in humans. Epidemiologic data indicate that it is an independent negative predictor for survival. If this is true in a controlled randomized study, it could be due to effects of the drug itself or more likely due to reduced quality of chest compressions and ventilations due to the time spent on placing an I.V. needle and injecting drugs.

DETAILED DESCRIPTION:
In a randomized, controlled study of all out-of-hospital cardiac arrest patients in Oslo, Norway, half the patients are treated according to the international guidelines for advanced CPR, and the other half according to the same guidelines, except for no I.V. needle or drugs are given until 5 minutes after eventual return of spontaneous circulation.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest out-of-hospital

Exclusion Criteria:

* <18 years old
* Trauma as cause of arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 904 (Actual)
Dates: Start 2003-01; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
survival to hospital discharge with neurologic outcome | discharge from hospital

SECONDARY OUTCOMES:
admit to hospital with spontaneous circulation | hospital admission
one year survival with neurologic outcome | one year after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wik, MD, PhD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Ulleval University Hospital, Oslo, Norway

REFERENCES:
- [Background] Holmberg M, Holmberg S, Herlitz J. Low chance of survival among patients requiring adrenaline (epinephrine) or intubation after out-of-hospital cardiac arrest in Sweden. Resuscitation. 2002 Jul;54(1):37-45. doi: 10.1016/s0300-9572(02)00048-5. PMID 12104107
- [Derived] Olasveengen TM, Sunde K, Brunborg C, Thowsen J, Steen PA, Wik L. Intravenous drug administration during out-of-hospital cardiac arrest: a randomized trial. JAMA. 2009 Nov 25;302(20):2222-9. doi: 10.1001/jama.2009.1729. PMID 19934423